CLINICAL TRIAL: NCT00689247
Title: A Phase I, Open, Randomised, Single-Centre, Crossover Study to Assess the Absorption, Distribution, Metabolism and Excretion (ADME) After Oral and Intravenous Administration of 14C-labelled and Non-labelled AZD1305 to Healthy Male Volunteers
Brief Title: To Study the Absorption, Distribution, Metabolism and Excretion of AZD1305
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Helen Lunde, MD, Medical Science Director, Emerging Arrhythmia and Lipids, AstraZeneca
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D3190C00008; 2007-007784-25 (EudraCT No)
Record Dates: First submitted 2008-05-30; First posted 2008-06-03 (Estimated); Last update posted 2010-12-03 (Estimated); Status verified 2010-12

CONDITIONS: Healthy
Keywords: AZD1305; ADME; pharmacokinetic; Absorption; distribution; metabolism; excretion
MeSH Terms: interventions — tert-butyl (2-(7-(2-(4-cyano-2-fluorophenoxy)ethyl)-9-oxa-3,7-diazabicyclo(3.3.1)non3-yl)ethyl)carbamate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): AZD1305 given as oral solution
  Interventions: Drug: AZD1305
- B (Experimental): AZD1305 given as iv infusion
  Interventions: Drug: AZD1305

INTERVENTIONS:
Drug: AZD1305 — oral solution, single dose
  Arms: A
Drug: AZD1305 — iv infusion, single dose
  Arms: B

SUMMARY:
The purpose of this study is to learn more about how AZD1305 is handled by the body, i.e the absorption, distribution, metabolism and excretion of AZD1305.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* A body mass index (BMI=weight/height2) of 19 to 30 kg/m2

Exclusion Criteria:

* Potassium outside normal reference values
* ECG findings outside normal range

Ages: 35 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2008-04; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic variables | During all dosing visits

SECONDARY OUTCOMES:
Adverse events, vital signs, ECG, laboratory variables and physical examination | During the study

CONTACTS AND LOCATIONS:
Overall Officials: Helen Lunde, MD, Study Director — AstraZeneca R&D, Mölndal, Sweden; Raj Chetty, MBBS, MD, Principal Investigator — AstraZeneca CPU Alderley Park, United Kingdom
Locations (1):
- Research Site, Macclesfield, Cheshire, United Kingdom